CLINICAL TRIAL: NCT07047560
Title: Liposomal Irinotecan (II) Fractionated Dosing Combined With 5-FU/LV (FOLFIRInali-3) and Bevacizumab in Second-line Treatment of Advanced Colorectal Cancer: A Single-arm, Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJFOLFIRInali-3
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Liposomal irinotecan; colorectal cancer; fractionated dosing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liposomal irinotecan (II) fractionated dosing combined with 5-FU/LV and bevacizumab (Experimental): Liposomal irinotecan (II): 30 mg/m² IV on D1 and D3, Q2W Fluorouracil (5-FU): Q2W
  * 400 mg/m² IV bolus on D1
  * Followed by 2400 mg/m² continuous IV infusion over 46-48 hours Leucovorin (LV): 400 mg/m² IV infusion on D1 Bevacizumab: 5 mg/kg IV infusion on D1, Q2W
  Interventions: Drug: fractionated liposomal irinotecan (II)-based combination chemotherapy (FOLFIRInali-3) plus bevacizumab (Bev)

INTERVENTIONS:
Drug: fractionated liposomal irinotecan (II)-based combination chemotherapy (FOLFIRInali-3) plus bevacizumab (Bev) — Liposomal irinotecan (II): 30 mg/m² IV on D1 and D3, Q2W; Fluorouracil (5-FU): Q2W;
  * 400 mg/m² IV bolus on D1
  * Followed by 2400 mg/m² continuous IV infusion over 46-48 hours Leucovorin (LV): 400 mg/m² IV infusion on D1 Bevacizumab: 5 mg/kg IV infusion on D1, Q2W.

SUMMARY:
This is an investigator-initiated, prospective, multicenter, single-arm phase II clinical study. It aims to evaluate the efficacy and safety of fractionated liposomal irinotecan (II)-based combination chemotherapy (FOLFIRInali-3) plus bevacizumab (Bev) as second-line treatment for advanced colorectal cancer, with the primary endpoint being objective response rate (ORR).

Eligible subjects will receive second-line treatment with the FOLFIRInali-3 （Liposomal irinotecan (II) fractionated dosing combined with 5-FU/LV） plus bevacizumab (Bev) 。Treatment will be discontinued upon occurrence of any of the following: Disease progression (radiologically confirmed)，intolerable toxicity (unmanageable after dose modification)， initiation of new antitumor therapy, withdrawal of informed consent or investigator's discretion (based on clinical judgment). Patients received regular and periodic reviews, with imaging evaluations every 6 weeks.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, multicenter, single-arm phase II clinical study. It aims to evaluate the efficacy and safety of fractionated liposomal irinotecan (II)-based combination chemotherapy (FOLFIRInali-3) plus bevacizumab (Bev) as second-line treatment for advanced colorectal cancer, with the primary endpoint being objective response rate (ORR).

Prospective participants must undergo screening assessments within 28 days before randomization to determine eligibility. Eligible subjects will receive second-line treatment with the FOLFIRInali-3 plus bevacizumab (Bev) regimen as follows:

1. Liposomal irinotecan (II): 30 mg/m² IV on D1 and D3
2. Fluorouracil (5-FU):

   * 400 mg/m² IV bolus on D1
   * Followed by 2400 mg/m² continuous IV infusion over 46-48 hours
3. Leucovorin (LV): 400 mg/m² IV infusion on D1
4. Bevacizumab: 5 mg/kg IV infusion on D1。

Treatment will be discontinued upon occurrence of any of the following:

1. Disease progression (radiologically confirmed)
2. Intolerable toxicity (unmanageable after dose modification)
3. Initiation of new antitumor therapy
4. Withdrawal of informed consent
5. Investigator's discretion (based on clinical judgment)

Patients received regular and periodic reviews, with imaging evaluations every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent；
2. Male or female patients ≥18 years old;
3. ECOG physical status score is 0 or 1;
4. Patients with pathologically confirmed advanced colorectal carcinoma (all other histological types excluded);
5. Patients who experienced disease progression under either of the following circumstances:During or within 6 months after first-line oxaliplatin-containing chemotherapy, or within 1 year after completing oxaliplatin-based adjuvant chemotherapy post-resection;
6. Expected survival time ≥ 3 months;
7. Patients must have at least one measurable metastatic lesion according to RECIST version 1.1;
8. Normal organ function:

   1. Hematology :Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/mm3); Platelet count ≥ 100 × 109/L (100000/mm3); Hemoglobin ≥ 90g/L;
   2. Kidney:The calculated value of creatinine clearance rate (CrCl) is ≥ 50 mL/min; Normal urine routine, urine protein<2+or 24-hour (h) urine protein quantification<1.0 g;
   3. Liver:Total serum bilirubin (TBiL) ≤ 1.5 × ULN;AST and ALT ≤ 2.5 × ULN; For subjects with liver metastasis, AST and ALT can be ≤ 5 × ULN;Serum albumin (ALB) ≥ 30g/L;
   4. Normal coagulation function, international standardized ratio (INR) ≤ 1.5 x ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
9. Women of childbearing age must undergo a pregnancy test (serum or urine) with a negative result within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug; For males, surgical sterilization or agreement to use appropriate methods of contraception during observation and within 8 weeks after the last administration of study medication should be considered;
10. Comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study;

Exclusion Criteria:

1. History of other malignancies (except cured basal cell carcinoma or cervical carcinoma in situ);
2. Participation in other drug trials within 4 weeks prior to enrollment;
3. Uncontrolled hypertension (SBP >160 mmHg or DBP >100 mmHg);
4. Acute coronary syndrome (including MI/unstable angina) with coronary angioplasty/stent placement within 6 months;
5. NYHA class II+ heart failure, unstable angina, MI, or severe arrhythmia with cardiovascular impairment within 6 months;
6. Symptomatic brain metastases;
7. Severe comorbidities requiring hospitalization (e.g., ileus, bowel obstruction, pulmonary fibrosis, refractory diabetes, heart/kidney/liver failure, psychiatric/cerebrovascular disorders);
8. Gastrointestinal perforation/fistula, intra-abdominal abscess, or non-GI fistula within 6 months;
9. Concomitant use of strong CYP3A4/CYP2C8 inhibitors/inducers or UGT1A1 inhibitors within 2 weeks;
10. Pregnancy or lactation;
11. Other investigator-determined contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate,ORR | 6 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival,OS | 24 months
  Defined as the time between signing the informed consent form to death due to various causes.
Incidence of adverse events | 24 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No